CLINICAL TRIAL: NCT06567548
Title: Clinical Comparison of Albumin Platelet Rich- Fibrin (Alb-PRF) Versus Platelet-rich Fibrin (PRF) on Postoperative Morbidity Following Free Gingival Graft Harvesting: a Randomized Controlled Clinical Trial
Brief Title: Clinical Comparison of Alb-PRF Vs PRF on Postoperative Morbidity Following FGG Harvesting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Samar Idris Hamelin Idris, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17624
Record Dates: First submitted 2024-08-19; First posted 2024-08-22 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Palate; Wound
Keywords: PRF; Alb-PRF; FGG
MeSH Terms: conditions — Wounds and Injuries | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): absorbable gelatin sponge
  Interventions: Other: control group
- Platelet-rich fibrin (PRF) group (Active Comparator): Platelet-rich fibrin (PRF) is a biomaterial derived from the patient's own blood, utilized primarily in regenerative medicine and surgery due to its rich content of growth factors and its ability to promote healing.
  Interventions: Other: Platelet-rich fibrin (PRF)
- Albumin Platelet Rich- Fibrin (Alb-PRF) group: (Experimental): Albumin Platelet-Rich Fibrin (Alb-PRF) is an innovative biomaterial that combines the regenerative properties of platelet-rich fibrin (PRF) with the structural and functional benefits of albumin. This mixture is designed to enhance tissue healing and regeneration by utilizing autologous blood components.
  Interventions: Other: Albumin Platelet Rich- Fibrin

INTERVENTIONS:
Other: control group — An absorbable gelatin sponge is a sterile hemostatic agent primarily composed of purified porcine-derived gelatin. It is widely utilized in surgical procedures to control bleeding
  Arms: Control group
Other: Platelet-rich fibrin (PRF) — Platelet-rich fibrin (PRF) is a biomaterial derived from the patient's own blood, utilized primarily in regenerative medicine and surgery due to its rich content of growth factors and its ability to promote healing.
  Arms: Platelet-rich fibrin (PRF) group
Other: Albumin Platelet Rich- Fibrin — is an innovative biomaterial that combines the regenerative properties of platelet-rich fibrin (PRF) with the structural and functional benefits of albumin. This mixture is designed to enhance tissue healing and regeneration by utilizing autologous blood components.
  Arms: Albumin Platelet Rich- Fibrin (Alb-PRF) group:

SUMMARY:
Clinical Comparison of Albumin Platelet Rich- Fibrin (Alb- PRF) versus Platelet-rich fibrin (PRF) on Postoperative Morbidity Following Free Gingival Graft Harvesting: A Randomized Controlled Clinical Trial(RCT)

Study settings:

* The study will be conducted in the Oral Medicine and Periodontology department, Faculty of Dentistry - Cairo University, Egypt.
* Patients will be selected from the Department of Oral Medicine and Periodontology-Cairo University outpatient clinic.

Expected Duration of Participation and Number of Participants: Research Duration: 28 days Number of Participants: 39 volunteers

Work Plan:

During the first visit, preoperative photographs will be taken. Then, participants will be randomly assigned (using a website) into three groups:

Group A: Application of Alb-PRF at the donor site of the free gingival graft. Group B: Application of PRF at the donor site of the free gingival graft. Control: Application of Gelatin Sponge at the donor site.

* 10 ml of venous blood will be drawn from the patient to prepare Alb-PRF and PRF membranes for placement at the donor site.
* The membrane or gelatin sponge will be placed at the donor site and sutured.

Postoperative Protocol:

After surgery, patients will be instructed to take 600 mg of ibuprofen, and 0.12% chlorhexidine gluconate mouthwash for two weeks postoperatively.

Analgesics will be recommended only if there is pain, and no antibiotics will be prescribed.

Patients will receive verbal and written dietary advice postoperatively. They will be encouraged to avoid heat sources and adhere to a diet of cold and soft foods.

Cleaning the adjacent palatal side of the surgical site will be prohibited to avoid irritation, while gentle cleaning will be recommended after dressing removal.

In case of postoperative problems such as unusual bleeding or gum recession, patients will be provided with contact information for their physician for early intervention.

During Visual Analog Scale (VAS) pain recording, patients will be instructed only to describe pain from the palate and to track additional analgesic intake and consumed tablets. Follow-up visits will be scheduled on days 3, 7, 14, 21, and 28 postoperatively.

Postoperative Follow-up:

Palatal sutures will be removed after 7 days post-surgery. On days 14, 21, and 28, wound healing, tissue color match, complete re-epithelialization of the wound, and clinical wound healing area will be monitored.

DETAILED DESCRIPTION:
General Operative Procedures: Preoperative Evaluation

* Intra-Oral Examination: Confirm the patient's eligibility based on predefined criteria.
* Phase I Therapy: Perform thorough supragingival scaling and subgingival debridement.
* Plaque Control: Ensure the patient maintains proper mechanical and chemical plaque control.

Clinical Procedure: Free Gingival Graft (FGG) Harvesting

* Preparation: All procedures will be done under sterile conditions and local anesthesia
* FGG Harvesting:
* FGG will be harvested from the palate).
* Make two horizontal incisions (coronal incision 2mm above the gingival margin) and two vertical incisions to outline the graft area.
* Insert a blade along the coronal incision, perpendicular to the bone, then move parallel to the hard palate in a mesiodistal direction to detach the graft while maintaining uniform thickness and avoiding the palatal periosteum.
* Place the graft on sterile saline gauze to prevent shrinkage.
* Control Group:
* Apply an absorbable gelatin sponge to the wound after FGG harvesting.
* Secure with compressive palatal sling sutures ( 5-0 polypropylene).
* PRF Group:
* PRF Preparation: Collect 10 ml of intravenous blood, and centrifuge at 3000 Rounds Per Minute (RPM) for 10 minutes. Extract the PRF clot and form a membrane.
* Apply the PRF membrane over the donor site and secure it with criss-cross sutures ( 5-0 polypropylene).
* Alb-PRF Group:
* Alb-PRF Preparation: Collect 10 ml of intravenous blood, and centrifuge at 700 RPM for 8 minutes. Heat the upper layer to 75°C for 10 minutes to form albumin gel, then cool.

Mix the albumin gel with liquid PRF to form Alb-PRF.

* Apply the Alb-PRF membrane over the donor site and secure it with criss-cross sutures ( 5-0 polypropylene).

Postsurgical Care

* Pain Management: Take Ibuprofen 600 mg as needed.
* Mouthwash: Use 0.12% chlorhexidine gluconate for two weeks.
* Dietary Instructions: Follow a cold, soft diet; avoid hot foods.
* Oral Hygiene: Avoid brushing near the surgical site; gentle brushing is allowed after pack removal.
* Emergency Contact: Provided for issues like abnormal bleeding.
* Pain Assessment: Use the Visual Analog Scale (VAS) to assess pain in the palate.
* Follow-Up: Scheduled for 3, 7, 14, 21, and 28 days post-surgery.
* Suture Removal: 7 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in need of free gingival graft
2. Medically free patients
3. Adult patients above 18 years old.
4. Patients accepting a 1-month follow-up period (cooperative patients).
5. Patients who will provide an informed consent.

Exclusion Criteria:

1. Smokers
2. Pregnant and lactating women
3. Patients with poor oral hygiene
4. Patients who had previous periodontal surgery in the area of interest

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain (PP) | VAS will be recorded daily for day 1, 3,7, and 14
  The patient will report their pain score directly through VAS score (between 0 and 10; 0: no pain, 1:
  minimal pain, 5: moderate pain, and 10: severe pain).

SECONDARY OUTCOMES:
Indirect postoperative pain | for 7 days postoperatively
  Will be assessed indirectly by mean consumption of analgesics
Tissue color match (TCM) | will be assessed on day 3, day 7, day 14, day 21, and day 28
  The palatal mucosa's color using Visual analog Scale,VAS Scale (0-10)
  Qualitative Ordinal (VAS
Complete wound re-epithelialization (CWE) | day 28
  Complete healing will be assessed using Bubbling test (yes or No) on day 28 and can be confirmed by applying hydrogen peroxide to the wound.
Wound clinical healing area | will be assessed on day 3, day 7, day 14, day 21, and day 28
  Measurement of wound closure area using University of North Carolina (UNC-15) periodontal probe to measure the size of palatal wound (width x length) and depth in millimeters.
Delayed wound bleeding (DWB) | day 7
  measuring the time of the Measuring the time of the bleeding (Hours, days, weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Enji Mahmoud, Phd, Study Director — Cairo University; Sarah Elbanna, Phd, Study Director — Cairo University
Locations (1):
- Cairo University, Cairo, Cairo Governorate, Egypt